CLINICAL TRIAL: NCT04071769
Title: Using Xenon MRI to Evaluate the Efficacy of Therapies for Idiopathic Pulmonary Fibrosis
Brief Title: Genentech Xenon MRI Idiopathic Pulmonary Fibrosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Principal Investigator, Bastiaan Driehuys, Professor of Medicine, Duke University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00101911
Record Dates: First submitted 2019-08-09; First posted 2019-08-28 (Actual); Results first posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Newly Diagnosed Idiopathic Pulmonary Fibrosis (IPF) (Experimental): Whether magnetic resonance imaging (MRI) using inhaled hyper-polarized 129 Xenon gas can help visualize impaired lung function to detect changes over time in Idiopathic Pulmonary Fibrosis (IPF) patients receiving approved IPF treatments
  Interventions: Drug: Hyperpolarized 129 Xenon Gas Comparing Idiopathic Pulmonary Fibrosis (IPF) Treatment

INTERVENTIONS:
Drug: Hyperpolarized 129 Xenon Gas Comparing Idiopathic Pulmonary Fibrosis (IPF) Treatment — Whether magnetic resonance imaging (MRI) using inhaled hyper-polarized 129 Xenon gas can help visualize impaired lung function to detect changes over time in Idiopathic Pulmonary Fibrosis (IPF) patients receiving approved IPF treatments

SUMMARY:
The purpose of this study is being done to determine whether magnetic resonance imaging (MRI) using inhaled hyper-polarized 129 Xenon gas can help visualize impaired lung function to detect changes over time in Idiopathic Pulmonary Fibrosis (IPF) patients receiving approved IPF treatments.

Participants will undergo an approximately hour long comprehensive MRI protocol, including administration of multiple doses of hyper-polarized 129 Xenon. The subjects will have this initial study prior to initiation of IPF therapies. Then the participants will have repeat studies at 3, 6 and 12 months following the initiation of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients of either gender, age > 18.
* Willing and able to give informed consent and adhere to visit/protocol schedules.

(Consent must be given before any study procedures are performed)

* Clinical diagnosis of IPF by confirmed by multidisciplinary diagnosis and naïve to treatment with an approved IPF therapy (either nintedanib or pirfenidone)

Exclusion Criteria:

* Subject is less than 18 years old
* Subjects who have been previously on either pirfenidone or nintedanib
* MRI is contraindicated based on responses to MRI screening questionnaire
* Subject is pregnant or lactating
* Resting oxygen saturation on room air <90% on supplemental oxygen
* Respiratory illness of a bacterial or viral etiology within 30 days of MRI
* Subject with ventricular cardiac arrhythmia in the past 30 days.
* Subject has history of cardiac arrest within the last year
* Subject does not fit into 129 Xenon vest coil used for MRI
* Subject deemed unlikely to be able to comply with instructions during imaging
* Recent exacerbation (within 30 days) defined by the need for antibiotics and/or systemic steroids
* Medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2029-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Tighe, MD, Principal Investigator — Duke University Health Systems
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Newly Diagnosed Idiopathic Pulmonary Fibrosis (IPF)
Started | 34
Completed | 21
Not Completed | 13
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Population: Participants who began treatment with antifibrotic.
Arm/Group | Newly Diagnosed Idiopathic Pulmonary Fibrosis (IPF)
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.56 (6.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Efficiency of Gas Exchange as Measured by the Red Blood Cell (RBC):Barrier Ratio Following Initiation of IPF Therapy
Description: RBC:barrier ratio will be determined using 129 Xenon MRI. The RBC:barrier ratio is a key metric that quantifies the efficiency of gas exchange, specifically the balance between red blood cell uptake and alveolar-capillary barrier function by showing how well oxygen gets from the air sacs to the blood. A low ratio often indicates impaired gas transfer, reflecting conditions where either RBC function or the barrier's permeability is compromised.
Time Frame: Baseline, 3, 6, and 12 months following initiation of IPF therapy
Measure: Mean (Standard Deviation); unit: RBC:barrier ratio
Arm/Group | Newly Diagnosed Idiopathic Pulmonary Fibrosis (IPF)
Number analyzed (Participants) | 25
RBC:barrier ratio
  Baseline | 0.250 (0.062)
  3 months | 0.237 (0.071)
  6 months | 0.246 (0.073)
  12 months | 0.256 (0.063)
Statistical Analysis 1: Comparison: Newly Diagnosed Idiopathic Pulmonary Fibrosis (IPF); Null hypothesis: there is no difference in the Xenon MRI measure of RBC-to-Membrane (RBC:M) at baseline vs. 3 months after initiating anti-fibrotic therapy; Test type: Other; p = 0.27, t-test, 2 sided

2. Secondary Outcome: Change in Pulmonary Function Following Initiation of IPF Therapy - Forced Vital Capacity (FVC)
Description: FVC, or Forced Vital Capacity, is a lung function test that measures the maximum amount of air a person can forcefully exhale from their lungs after taking a deep breath. This test is performed using a spirometer and the results are used by healthcare providers to help diagnose and monitor pulmonary diseases like asthma, emphysema, or restrictive lung conditions.
Time Frame: Baseline, 3, 6, and 12 months following initiation of IPF therapy
Population: Two participants only completed the baseline visit.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Newly Diagnosed Idiopathic Pulmonary Fibrosis (IPF)
Number analyzed (Participants) | 23
liters
  Baseline to 3 months | 0.073 (0.244)
  Baseline to 6 months | 0.063 (0.229)
  Baseline to 12 months | 0.190 (0.256)
Statistical Analysis 1: Comparison: Newly Diagnosed Idiopathic Pulmonary Fibrosis (IPF); Test type: Other — Baseline to 3 months; p = 0.23, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Newly Diagnosed Idiopathic Pulmonary Fibrosis (IPF); Test type: Other — Baseline to 6 months; p = 0.26, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Newly Diagnosed Idiopathic Pulmonary Fibrosis (IPF); Test type: Other — Baseline to 12 months; p = 0.68, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Pulmonary Function Following Initiation of IPF Therapy - Diffusion Capacity for Carbon Monoxide (DLCO)
Description: The DLCO, or Diffusing Capacity of the Lung for Carbon Monoxide, is a pulmonary function test that measures how well oxygen transfers from the lungs to the blood by measuring how much carbon monoxide diffuses from the lungs into the bloodstream. Performed by inhaling a special gas mixture and holding the breath, the DLCO test assesses the gas exchange function of the lungs.
Time Frame: Baseline, 3, 6, and 12 months following initiation of IPF therapy
Population: Participants with data collected at both timepoints used for analysis. Two participants only completed the baseline visit.
Measure: Mean (Standard Deviation); unit: mL/min/mmHg
Arm/Group | Newly Diagnosed Idiopathic Pulmonary Fibrosis (IPF)
Number analyzed (Participants) | 22
mL/min/mmHg
  Baseline to 3 months | 0.026 (1.961)
  Baseline to 6 months: number analyzed (Participants) | 19
  Baseline to 6 months | -0.029 (2.530)
  Baseline to 12 months: number analyzed (Participants) | 20
  Baseline to 12 months | -0.306 (1.846)
Statistical Analysis 1: Comparison: Newly Diagnosed Idiopathic Pulmonary Fibrosis (IPF); Test type: Other — Baseline to 3 months; p = 0.95, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Newly Diagnosed Idiopathic Pulmonary Fibrosis (IPF); Test type: Other — Baseline to 6 months; p = 0.92, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Newly Diagnosed Idiopathic Pulmonary Fibrosis (IPF); Test type: Other — Baseline to 12 months; p = 0.56, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Up to 18 months
Arm/Group | Newly Diagnosed Idiopathic Pulmonary Fibrosis (IPF)
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT04071769/Prot_SAP_000.pdf